CLINICAL TRIAL: NCT06859606
Title: Mandibular Sequential Distalization Versus Class III Elastics With Clear Aligners in Class III Patients: a Randomized Controlled Trial
Brief Title: Mandibular Sequential Distalization Versus Class III Elastics With Clear Aligners in Class III Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Camillus International University of Health Sciences (Other)
Responsible Party: Principal Investigator, Francesca Gazzani, Research Assistant, Saint Camillus International University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 75.23
Record Dates: First submitted 2025-02-11; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Class III Malocclusion
Keywords: class III malocclusion; lower molar distalization; class III elastics; clear aligner treatment
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Lower Distalization Protocol (Experimental): In Group 1 (Lower Distalization Protocol), all subjects underwent lower molar distalization combined with Class III elastics.
  Interventions: Other: Lower molar distalization
- Group 2, Non-Distalization Protocol (Experimental): In Group 2 (Non-Distalization Protocol) all subjects were treated with dento-alveolar expansion and Class III elastics
  Interventions: Other: Class III elastics

INTERVENTIONS:
Other: Lower molar distalization — Lower Distalization Protocol included extraction of the lower third molars before starting treatment and a 50% sequential lower distalization with two teeth being distalized at a time. The distalization started with the movement of lower second molars, followed by the first molars halfway through the process, and so on. Once the canine reached the right position, the "en masse" retraction of the four incisors completed the treatment plan. The protocol comprised the use of Class III intermaxillary elastics to support the distalization movement and to control the proclination of lower incisors
  Arms: Group 1 - Lower Distalization Protocol
Other: Class III elastics — Non-Distalization Protocol featured extraction of the lower third molars before starting treatment, transversal dento-alveolar coordination, strategic interproximal reduction (IPR) in the anterior segment of the lower arch, and the addition of Class III elastics
  Arms: Group 2, Non-Distalization Protocol

SUMMARY:
Distalizing mandibular molars may be indicated for patients with minor skeletal Class III discrepancies or in Class III subjects with mild crowding. Traditionally, mandibular molar distalization was accomplished using elastics, open coils, and the multiloop edgewise archwire technique. In recent years, several techniques have been developed to reduce the dependence on patient compliance, such as skeletal anchorage. Recently, several reports have been published on mandibular distal movement using miniscrews and some case reports have shown the possibility of obtaining Class III correction with sequential mandibular distalization in non-growing subjects by means of clear aligners. However, a sound clinical judgment should always be made on the basis of a higher level of evidence. Therefore, the purpose of the present prospective study is to provide a detailed analysis of the underlying skeletal and dental changes determined by mandibular distalization therapy with the sequential Invisalign protocol in permanent dentition. This will be accomplished by testing the following null hypothesis: mandibular molar distalization is not achievable with aligners without the application of TADs.

DETAILED DESCRIPTION:
Class III malocclusion is considered one of the most challenging maxillofacial disorders in clinical practice characterized by an antero-posterior discrepancy with mandibular protrusion, maxillary retrusion, or a combination of both. In adult patients, managing this condition is further complicated by the absence of residual skeletal growth, limiting therapeutic options to orthodontic interventions and, in some cases, surgical procedures. Diagnosis in Class III adult patients requires distinguishing between skeletal malocclusion and dento-alveolar discrepancy. The combination of orthognathic surgery and orthodontic therapy represents the gold standard for more severe skeletal Class III disharmonies, leading to an improvement of both function and aesthetics. On the other hand, in Class III cases characterized by a prevalent dental component or mild skeletal discrepancy, the malocclusion can be addressed with a dento-alveolar compensation. In these cases, the clinical objectives are to achieve a correct sagittal, canine and molar Class I relationship, as well as ideal values of overjet and overbite. The non-surgical orthopedic approach involves the application of Class III elastics or the distalization of the lower molars, which can improve the sagittal occlusal relationship. As a matter of fact, mandibular distalization allows the increase of lower arch length along with the achievement of the necessary space to correct a Class III relationship. However, bone density and root anatomy make lower molar distalization difficult to achieve. In addition, one of the most frequent adverse effects is represented by the anterior anchorage loss with a worsening of lower incisor proclination and overjet values. Traditional appliances feature the use of open coil springs, inter arch elastics, and lip bumper device combined with fixed appliances. Nowadays, the development of clear aligner technology provides new opportunities even in the management of complex malocclusion cases, including Class III discrepancies. In particular, molar distalization movements and intermaxillary elastics have been proposed as a valid clinical strategy to improve the occlusal relationship without requiring skeletal anchorage devices. During the sagittal mechanics, over-corrected movements should be planned in order to obtain more bodily movements of the lower molars. Moreover, the best accuracy and predictability of distalization movements are supported by the sequential staging and the presence of attachments on the tooth surfaces. Nowadays, scientific evidence on this topic is limited and it is influenced by restrictions in terms of sample size, retrospective design, and lack of long-term observation. Hence, the aim of the present study was to evaluate the efficacy and efficiency of intermaxillary elastics combined with lower molar distalization by means of clear aligners in the treatment of Class III malocclusion in adult patients. More specifically, a randomized controlled trial (RCT) was conducted to evaluate the antero-posterior correction induced by Class III elastics combined with lower distalization movements and the application of Class III elastics alone. The possibility of achieving satisfying clinical outcomes without the use of skeletal anchorage was considered to avoid an invasive orthodontic approach

ELIGIBILITY:
Inclusion Criteria:

* adult age (≥19 years)
* permanent dentition including second permanent molars
* skeletal Class I or slight Class III (-2° < ANB < +2°)
* normal skeletal divergency pattern (SN^GoGn, 27°-37°)
* Class III canine and molar relationship at baseline (T0), moderate lower arch crowding (≤ +4 mm)
* good compliance with aligners and elastics (≥ 20 hours/day)

Exclusion Criteria:

* severe skeletal Class III malocclusion (ANB < -2°)
* transversal maxillary deficiency
* use of Temporary Anchorage Devices (TADs)
* extraction treatments other than third molars
* periodontal disease or temporomandibular disorders (TMDs).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Lower molar positional changes expressed by means of linear and angular measurements (L6-MP mm; L6-MP angle; L6 - CoGo mm; L6 apex - CoGo mm) | from the start of treatment to the end at 24 months
  L6-MP mm: linear distance between the mesial cusp of lower first molar and Mandibular plane L6-MP angle: angle between long axis of lower first molar and Mandibular plane L6 - CoGo mm: linear distance between the mesial cusp of lower first molar and CoGo line L6 apex - CoGo mm: linear distance between the apex of lower first molar and CoGo line

SECONDARY OUTCOMES:
Changes in inclination of the lower incisors (IMPA angle) | from the start of treatment to the and at 24 months
  IMPA angle: angle between long axis of the lower incisor and mandibular plane
Changes in position of the lower incisors (L1-CoGo mm; L1apex - CoGo) | from the start of treatment to the and at 24 months
  L1-CoGo mm: linear distance between the tip crown of the lower incisor L1apex - CoGo mm: linear distance between the apex of the lower incisor and CoGo line
Sagittal skeletal changes (SNA angle, SNB angle, ANB angle) | from start of treatment to to the end at 24 months
  SNA angle: maxillary sagittal position SNB angle: mandibular sagittal position ANB angle: maxillomandibular sagittal discrepancy
Sagittal skeletal changes (Wits appraisal) | from start of treatment to to the end at 24 months
  Wits appraisal: maxillomandibular sagittal discrepancy
Vertical skeletal changes (SN^MP angle, Gonial Angle) | from the start of treatment to the end at 24 months
  SN-MP angle between Sella/Nasion plane and Mandibular plane Gonial angle, angle between Ar-Go plane and Go-Me plane
Changes of upper incisors inclination | from the start of treatment to the and at 24 months
  Incisor inclintion: angle between long axis of upper incisor and Sella Nasion
Overbite and Overjet values | from the start of treatment to the and at 24 months
  Overbite mm: horizontal distance between the upper and lower incisors on the occlusal plane Overjet mm: vertical distance between the upper and lower incisors on the occlusal plane

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Camillus International University of Health Sciences, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martina H, Stefano Adriana A, Ernesto B, Alessandra I, Roberto AV, Gabriella G. Lower molar distalization using clear aligners: Is it effective? A systematic review. J Orthod Sci. 2024 Feb 16;13:11. doi: 10.4103/jos.jos_174_23. eCollection 2024. PMID 38516119
- [Background] Rota E, Parrini S, Malekian K, Cugliari G, Mampieri G, Deregibus A, Castroflorio T. Lower molar distalization using clear aligners: bodily movement or uprighting? A preliminary study. Appl. Sci. 2022, 12(14), 7123.
- [Background] Han J, Ning N, Du H, Zhou M, Cai C, Hong Y, et al. Efficacy of clear aligners on mandibular molar distalization: A retrospective study. Digit Med 2021; 7:1.
- [Background] Padmanabhan A, Khan Y, Lambate V, K U, Naveed N, Singh M, Nagi PK. Efficacy of Clear Aligners in Treating Class III Malocclusion With Mandibular Molar Distalization: A Systematic Review. Cureus. 2023 Nov 1;15(11):e48134. doi: 10.7759/cureus.48134. eCollection 2023 Nov. PMID 38046776
- [Background] Pavoni C, Gazzani F, Franchi L, Loberto S, Lione R, Cozza P. Soft tissue facial profile in Class III malocclusion: long-term post-pubertal effects produced by the Face Mask Protocol. Eur J Orthod. 2019 Sep 21;41(5):531-536. doi: 10.1093/ejo/cjz003. PMID 30865768
- [Derived] Gazzani F, Pavoni C, De Razza FC, Lugli L, Cozza P, Lione R. Clear aligner treatment in adult patients with class III malocclusion: lower distalization and class III elastics vs class III elastics alone - a RCT. Eur J Orthod. 2025 Jun 12;47(4):cjaf052. doi: 10.1093/ejo/cjaf052. PMID 40600239